CLINICAL TRIAL: NCT00259207
Title: Pulmonary Valve Replacement : Study of Comparison Between a Standard Surgical Approach With Extracorporeal Circulation and an Off-pump Hybrid Strategy.
Brief Title: Pulmonary Valve Replacement in Large Right Ventricular Outflow Tract
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other); European Georges Pompidou Hospital (Other)
Responsible Party: Cecile Jourdain, Department Clinical Research of Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040413; AOR04068
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2007-03

CONDITIONS: Pulmonary Valve Insufficiency
Keywords: Pulmonary valve regurgitation; Valve replacement; Hybrid procedure
MeSH Terms: conditions — Pulmonary Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- classic surgery (Active Comparator): classic surgery
  Interventions: Procedure: Pulmonary valve insertion
- medical surgery hybride (Experimental): medical surgery hybride
  Interventions: Procedure: medical surgery hybride

INTERVENTIONS:
Procedure: Pulmonary valve insertion — Pulmonary valve insertion
  Arms: classic surgery
Procedure: medical surgery hybride — medical surgery hybride
  Arms: medical surgery hybride

SUMMARY:
The purpose of this study is to compare 2 techniques of pulmonary valve replacement in patients with a large right ventricular outflow tract: a standard surgical treatment using cardiopulmonary bypass versus a medico-surgical hybrid strategy without extracorporeal circulation.

DETAILED DESCRIPTION:
Pulmonary regurgitation is a common complication late after complete correction of a tetralogy of Fallot. It progressively leads to a right ventricular dilatation that has been strongly associated with ventricular arrhythmia, sudden death and right ventricular insufficiency. Pulmonary valve replacement reduces the rate of complications but the precise timing for this procedure remains unknown. Moreover, pulmonary valve replacement, even before the occurrence of symptoms, doesn't allow for a total recovery in all patients. Reasons are not known, but cardiopulmonary bypass as well as late referral to surgery have been incriminated to explain the persistence of right ventricular dysfunction after surgical valvular. Therefore, a strategy avoiding cardiopulmonary bypass could potentially preserve the right ventricular function and in the meantime reduce the hospitalisation length and morbid-mortality. For the last six years, we and others have developed a technique of percutaneous pulmonary valve implantation. Encouraging results were reported in the treatment of failing right ventricular to pulmonary artery conduit, but presents indications are limited and the innovative technique could not be offered to most of patients requiring pulmonary valve replacement. In particular, to date, conventional surgery is the only approach for patients with large pulmonary trunk over 22 mm in diameter. We had the idea of collaborating with the surgeons to try to improve the outcome of valvular in these patients. We would like to investigate a hybrid strategy in those patients with large right ventricular outflow tract inaccessible to solely transcatheter technique. The studied technique will associate a surgical pulmonary artery banding without cardiopulmonary bypass immediately followed by a transventricular or a transvenous pulmonary valve insertion using a conventional valved stent. The purpose of this randomized study is to evaluate benefits and risks of the medico-surgical hybrid strategy, and to compare both strategies hybrid approach and conventional surgery with extracorporeal circulation in term of right ventricular function recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with surgical indication of pulmonary valve replacement for significant pulmonary regurgitation
2. Pulmonary trunk diameter > 22mm
3. Age > 5 years old or weight > 20kg
4. Acceptance of protocol
5. Social regimen security

Exclusion Criteria:

1. No indication of pulmonary valve replacement
2. Age < 5 years old or weight < 20kg
3. Extra-cardiac disease with a vital prognosis under 6 months
4. Heparin and contrast allergy
5. Clinical or biological signs of infection
6. Pregnancy
7. Patients in emergency state
8. Patients included in an another research protocol during the last months

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Right ventricular function | during the study

SECONDARY OUTCOMES:
Morbidity and mortality | during the study
Length of stay | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Younes BOUDJEMLINE, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- NECKER HOSPITAL for Sick Children, 149 R. de SEVRES, Paris, France

REFERENCES:
- [Background] Boudjemline Y, Schievano S, Bonnet C, Coats L, Agnoletti G, Khambadkone S, Bonnet D, Deanfield J, Sidi D, Bonhoeffer P. Off-pump replacement of the pulmonary valve in large right ventricular outflow tracts: a hybrid approach. J Thorac Cardiovasc Surg. 2005 Apr;129(4):831-7. doi: 10.1016/j.jtcvs.2004.10.027. PMID 15821651